CLINICAL TRIAL: NCT00005080
Title: A Phase II Study of 506U78 in Patients With Previously Systemically Untreated Cutaneous T-cell Lymphoma (CTCL) or With Refractory or Relapsed Non-cutaneous Peripheral T-cell Lymphoma (PTCL)
Brief Title: 506U78 in Treating Patients With Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02324; CALGB-59901; U10CA031946 (NIH); CDR0000067687 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-04-06; First posted 2004-04-19 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Small Intestine Lymphoma; Stage I Cutaneous T-cell Non-Hodgkin Lymphoma; Stage I Mycosis Fungoides/Sezary Syndrome; Stage II Cutaneous T-cell Non-Hodgkin Lymphoma; Stage II Mycosis Fungoides/Sezary Syndrome; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Mycosis Fungoides/Sezary Syndrome; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — nelarabine

ARMS (1):
- Nelarabine (Experimental): Patients receive 506U78 IV over 2 hours on days 1, 3, and 5. Treatment repeats every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity. Patients achieving complete response receive up to 8 courses of therapy.
  Interventions: Drug: nelarabine

INTERVENTIONS:
Drug: nelarabine — Given IV
  Other Names: 506U78; Arranon; GW506U78

SUMMARY:
Phase II trial to study the effectiveness of 506U78 in treating patients who have lymphoma that has not been treated previously or that has not responded to previous treatment. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the complete and partial remission rates and remission duration in patients with cutaneous T-cell lymphoma or refractory or relapsed noncutaneous peripheral T-cell lymphoma treated with 506U78.

II. Determine the safety and toxicity of this treatment regimen in this patient population.

OUTLINE:

Patients receive 506U78 IV over 2 hours on days 1, 3, and 5. Treatment repeats every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity. Patients achieving complete response receive up to 8 courses of therapy.

Patients are followed every 3 months for 1 year and then every 6 months for 1 year or until relapse.

PROJECTED ACCRUAL: A total of 34-74 patients will be accrued for this study within 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented cutaneous T-cell lymphoma (CTCL) or noncutaneous peripheral T-cell lymphoma (PTCL) (needle aspirate or core biopsy of tissue or marrow as the sole means of diagnosis is not acceptable), confirmed by immunophenotyping, including:

  * Mycosis fungoides/Sezary syndrome
  * Peripheral T-Cell lymphomas (medium, mixed medium-large, large cell)
  * Variants of peripheral T-Cell lymphoma
  * Angioimmunoblastic T-Cell lymphoma (AILD); angiocentric lymphoma; intestinal T-Cell Lymphoma; adult T-Cell lymphoma/leukemia (ATLL); anaplastic Large Cell (CD30+) lymphoma, T-cell type Failure to submit pathology slides within 60 days of patient registration will result in patient being declared ineligible; Note: patients diagnosed more than one year prior to entry on this protocol must have a repeat lymph node biopsy. In the event of rapid tumor growth, rising LDH, or the onset of B symptoms in a period of time less than one year a rebiopsy is also required
* Biopsy and immunophenotyping should be performed to document relapse after prior treatment
* CTCL patients may have received one prior course of single-agent systemic chemotherapy for CTCL, but may not have received a multi-agent chemotherapy regimen; patients may have received prior local, topical, radiation- or electron beam-based, or chemotherapy-based treatment; examples of the latter would include, but not be limited to, cytokines such as interferon, retinoids, monoclonal antibodies, and fusion toxins
* PTCL patients may have failed only one or two prior treatment regimens (one of which may include peripheral stem cell transplantation)
* Patients must have measurable disease; patients with CTCL must have skin lesions which are measurable; whenever CT is specified, it should be understood that MRI may be substituted as long as the measurements for tumor response are made on two successive studies employing the same procedure

  * The following lesions are not considered measurable:

    * Barium studies
    * Ascites or pleural effusion
    * Bony disease (lesions if present should be noted)
    * Bone marrow
* No CNS lymphoma requiring intrathecal or craniospinal radiation therapy
* No history of a seizure disorder or grade 3 neurologic toxicity during prior treatment of lymphoma. Baseline neurologic status of all eligible patients is to be carefully recorded (particularly in elderly patients and those with conditions potentially predisposed to neurotoxicity, such as diabetes mellitus and prior exposure to neurotoxic agents); patients with prior neurologic dysfunction or toxicity from any cause must have recovered to grade 1 neurologic toxicity/dysfunction
* Performance status 0-2
* No known HIV disease; patients with a history of intravenous drug abuse or any other behavior associated with an increased risk of HIV infection should be tested for exposure to the HIV virus; patients who test positive or who are known to be infected are not eligible; an HIV test is not required for entry on protocol, but is required if the patient is perceived to be at risk
* Calculated Creatinine Clearance >= 50 ml/min

  * Unless attributable to lymphoma
  * To be calculated by method of Cockcroft-Gault
* Bilirubin >= 1.5 x upper limit of normal

  * Patients with hepatic dysfunction should enroll on CALGB 69803

Max Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2000-05; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Remission rate (complete and partial remission) | Up to 2 years
Remission duration | From the time of first reported complete or partial response (later confirmed) until time of documented relapse, assessed up to 2 years
  Remission duration will be estimated using the method of Kaplan Meier.
Toxicity as assessed by the NCI Common Toxicity Criteria (CTC) version 2.0 | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Myron Czuczman, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States